CLINICAL TRIAL: NCT03456076
Title: A Phase III, Open-Label, Randomized Study to Evaluate the Efficacy and Safety of Adjuvant Alectinib Versus Adjuvant Platinum-Based Chemotherapy in Patients With Completely Resected Stage IB (Tumors Equal to or Larger Than 4cm) to Stage IIIA Anaplastic Lymphoma Kinase Positive Non-Small Cell Lung Cancer
Brief Title: A Study Comparing Adjuvant Alectinib Versus Adjuvant Platinum-Based Chemotherapy in Patients With ALK Positive Non-Small Cell Lung Cancer
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BO40336; 2017-004331-37 (EudraCT Number)
Record Dates: First submitted 2018-03-06; First posted 2018-03-07 (Actual); Results first posted 2024-08-26 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Carcinoma, Non-Small-Cell Lung
Keywords: NSCLC, alectinib, ALK positive,adjuvant treatment, platinum based chemotherapy, complete resection, Stage IB-IIIA.
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — alectinib; Cisplatin; Vinorelbine; Gemcitabine; Pemetrexed; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Alectinib (Experimental)
  Interventions: Drug: Alectnib
- Platinum-Based Chemotherapy (Active Comparator)
  Interventions: Drug: Cisplatin; Drug: Vinorelbine; Drug: Gemcitabine; Drug: Pemetrexed; Drug: Carboplatin

INTERVENTIONS:
Drug: Alectnib — Participants will receive alectinib 600 mg orally BID until completion of treatment period (24 months) or recurrence of disease , unacceptable toxicity, withdrawal of consent or death, whichever occurs first.
  Other Names: RO5424802
  Arms: Alectinib
Drug: Cisplatin — Participants will receive Cisplatin 75 milligrams per square meter (mg/m^2) on Day 1 every 21 days IV intravenously (IV) until completion of treatment period (4 cycles), recurrence of disease, unacceptable toxicity, withdrawal of consent, or death, whichever occurs first."
  Arms: Platinum-Based Chemotherapy
Drug: Vinorelbine — Participants will receive Vinorelbine 25 mg/m^2 IV on Days 1 and 8 Q21D until completion of treatment period (4 cycles), recurrence of disease, unacceptable toxicity, withdrawal of consent, or death, whichever occurs first.
  Other Names: Navelbine
  Arms: Platinum-Based Chemotherapy
Drug: Gemcitabine — Participants will receive Gemcitabine 1250 mg/m^2 on Days 1 and 8 Q21D IV until completion of treatment period (4 cycles), recurrence of disease, unacceptable toxicity, withdrawal of consent, or death, whichever occurs first.
  Other Names: Gitrabin
  Arms: Platinum-Based Chemotherapy
Drug: Pemetrexed — Participants will receive 500 mg/m^2 Day 1 Q21D until completion of treatment period (4 cycles), recurrence of disease, unacceptable toxicity, withdrawal of consent, or death, whichever occurs first."
  Other Names: Alimta®
  Arms: Platinum-Based Chemotherapy
Drug: Carboplatin — For participants who experience unacceptable toxicity with cisplatin, carboplatin can be used.
  Arms: Platinum-Based Chemotherapy

SUMMARY:
This randomized, active-controlled, multicenter, open-label, Phase III study is designed to investigate the efficacy and safety of alectinib compared with platinum-based in the adjuvant setting. Participants in the experimental arm will receive alectinib at 600 mg orally twice daily (BID) taken with food for 24 months.

Participants in the control arm will receive one of the protocol specified platinum based chemotherapy regimens for 4 cycles. Following treatment completion, participants will be followed up for their disease until disease recurrence. At the time of disease recurrence, participants will enter a survival follow-up until death, withdrawal of consent or study closure, whichever occurs earlier.

ELIGIBILITY:
Key Inclusion Criteria

* Age ≥18 years
* Complete resection of histologically confirmed Stage IB (tumor ≥ 4 cm) to Stage IIIA (T2-3 N0, T1-3 N1, T1-3 N2, T4 N0-1) NSCLC as per Union Internationale Contre le Cancer / American Joint Committee on Cancer, 7th edition, with negative margins, at 4-12 weeks before enrollment
* If mediastinoscopy was not performed preoperatively, it is expected that, at a minimum, mediastinal lymph node systematic sampling will have occurred
* Documented ALK-positive disease according to an FDA-approved and CE-marked test
* Eligible to receive a platinum-based chemotherapy regimen according to the local labels or guidelines
* Eastern Cooperative Oncology Group Performance Status of Grade 0 or 1
* Adequate hematologic and renal function
* For women of childbearing potential: agreement to remain abstinent or use contraceptive methods with a failure rate of < 1% per year during the treatment period and for at least 90 days after the last dose of alectinib or according to local labels or guidelines for chemotherapy
* For men: agreement to remain abstinent or use contraceptive measures, and agreement to refrain from donating sperm for at least 90 days after the last dose of alectinib or according to local labels or guidelines for chemotherapy. Men must refrain from donating sperm during this same period
* Willingness and ability to comply with scheduled visits, treatment plans, laboratory tests, and other study procedures

Key Exclusion Criteria

* Pregnant or breastfeeding, or intending to become pregnant during the study or within 90 days after the last dose of alectinib or according to local labels or guidelines for chemotherapy
* Prior adjuvant radiotherapy for NSCLC
* Prior exposure to systemic anti-cancer therapy and ALK inhibitors
* Stage IIIA N2 patients that, in the investigator's opinion, should receive post-operative radiotherapy treatment are excluded from the study
* Known sensitivity to any component of study drug to which the patient may be randomized. This includes, but is not limited to, patients with galactose intolerance, a congenital lactase deficiency or glucose-galactose malabsorption.
* Malignancies other than NSCLC within 5 years prior to enrollment, except for curatively treated basal cell carcinoma of the skin, early gastrointestinal (GI) cancer by endoscopic resection, in situ carcinoma of the cervix, ductal carcinoma in situ, papillary thyroid cancer, or any cured cancer that is considered to have no impact on disease free survival or overall survival for the current NSCLC
* Any GI disorder that may affect absorption of oral medications, such as malabsorption syndrome or status post-major bowel resection
* Liver disease characterized by aspartate transaminase and alanine transaminase >= 3 × upper limit of normal or impaired excretory function or synthetic function or other conditions of decompensated liver disease such as coagulopathy, hepatic encephalopathy, hypoalbuminemia, ascites, or bleeding from esophageal varices or active viral or active autoimmune, alcoholic, or other types of acute hepatitis
* Japanese patients participating in the serial/intensive PK sample collection only: administration of strong/potent CYP450 3A inhibitors or inducers within 14 days prior to the first dose of study treatment and while on treatment with alectinib up to Week 3
* Any exclusion criteria based on the local labels or guidelines for chemotherapy regimen
* Patients with symptomatic bradycardia
* History of organ transplant
* Known HIV positivity or AIDS-related illness
* Any clinically significant concomitant disease or condition that could interfere with-or for which the treatment might interfere with the conduct of the study or the absorption of oral medications or that would pose an unacceptable risk to the patients in this study, in the opinion of the Principal Investigator
* Any psychological, familial, sociological, or geographical condition potentially hampering compliance with the study protocol requirements and/or follow-up procedures; those conditions should be discussed with the patient before trial entry

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 257 (Actual)
Dates: Start 2018-08-16 (Actual); Primary Completion 2023-06-26 (Actual); Study Completion 2026-11-19 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (114):
- United States (3):
  - Rush University Medical Center, Chicago, Illinois
  - MGH Cancer Center, Boston, Massachusetts
  - AHN Cancer Institute ? Allegheny General Hospital, Pittsburgh, Pennsylvania
- Australia (3):
  - Chris O'Brien Lifehouse, Camperdown, New South Wales
  - GenesisCare North Shore, St Leonards, New South Wales
  - Peter MacCallum Cancer Center, Melbourne, Victoria
- Krankenhaus Nord - Klinik Floridsdorf, Vienna, Austria
- Belarus (3):
  - Healthcare Institution Grodno University Hospital, Hrodna, Grodnenskaya
  - Healthcare Institution ?Gomel Regional Clinical Oncologic Dispensary?, Homyel, Homyel'skaya Voblasts'
  - Vitebsk Regional Clinical Oncology Dispensary, Vitebsk, Vitebsk Oblast
- Clinical center University of Sarajevo, Sarajevo, Bosnia and Herzegovina
- China (12):
  - Beijing Cancer Hospital, Beijing
  - Jilin Cancer Hospital, Changchun
  - West China Hospital, Sichuan University, Chengdu
  - Fujian Medical University Union Hospital, Fujian
  - Guangdong General Hospital, Guangzhou
  - Zhejiang Cancer Hospital, Hangzhou
  - Shandong Cancer Hospital, Jinan
  - Shanghai Chest Hospital, Shanghai
  - Zhongshan Hospital Fudan University, Shanghai
  - Shenzhen People's Hospital, Shenzhen
  - Union Hospital Tongji Medical College Huazhong University of Science and Technology, Wuhan
  - First Affiliated Hospital of Medical College of Xi'an Jiaotong University, Xi'an
- Odense Universitetshospital, Onkologisk Afdeling R, Odense C, Denmark
- Kasr Eieny Uni Hospital, Cairo, Egypt
- France (4):
  - CHU Angers, Angers
  - Hopital Nord AP-HM, Marseille
  - Hopital Bichat Claude Bernard, Paris
  - Institut Gustave Roussy, Villejuif
- Germany (4):
  - Klinikum Chemnitz gGmbH, Chemnitz
  - Niels-Stensen-Kliniken Franziskus-Hospital Harderberg GmbH, Georgsmarienhütte
  - Thoraxklinik Heidelberg gGmbH, Heidelberg
  - Fachklinik für Lungenerkrankungen, Immenhausen
- Greece (2):
  - Metropolitan Hospital, Athens
  - Theageneio Hospital, Thessaloniki
- Hungary (2):
  - Orszagos Onkologiai Intezet, Budapest
  - Hetenyi Geza County Hospital, Szolnok
- Israel (2):
  - Rambam Health Care Campus, Haifa
  - Meir Medical Center, Kfar Saba
- Italy (5):
  - Az. Osp. Monaldi, Napoli, Campania
  - Azienda Ospedaliera San Camillo Forlanini - Unità Operativa Complessa di Pneumologia Oncologica 1, Rome, Lazio
  - Irccs Istituto Europeo di Oncologia (IEO), Milan, Lombardy
  - Azienda Ospedaliero-Universitaria San Luigi Gonzaga, Orbassano, Piedmont
  - Azienda Ospedaliera Di Perugia Ospedale s. Maria Della Misericordia, Perugia, Umbria
- Japan (18):
  - Aichi Cancer Center, Aichi
  - National Cancer Center Hospital East, Chiba
  - National Hospital Organization Kyushu Cancer Center, Fukuoka
  - Hiroshima University Hospital, Hiroshima
  - National Hospital Organization Hokkaido Cancer Center, Hokkaido
  - National Hospital Organization Himeji Medical Center, Hyōgo
  - Kanagawa Cancer Center, Kanagawa
  - Kumamoto University Hospital, Kumamoto
  - Kyoto University Hospital, Kyoto
  - Sendai Kousei Hospital, Miyagi
  - Niigata Cancer Center Hospital, Niigata
  - Okayama University Hospital, Okayama
  - Osaka City General Hospital, Osaka
  - Shizuoka Cancer Center, Shizuoka
  - National Cancer Center Hospital, Tokyo
  - Juntendo University Hospital, Tokyo
  - The Cancer Institute Hospital of JFCR, Tokyo
  - Tokyo Medical University Hospital, Tokyo
- Almaty Oncology Center, Almaty, Kazakhstan
- North Macedonia (2):
  - PHI University Clinic of Radiotherapy and Oncology; Malignant diseases of thorax, Skopje
  - Private Health Organization Acibadem Sistina Hospital, Skopje
- Poland (4):
  - Gdanski Uniwersytet Medyczny, Gda?sk
  - Krakowski Szpital Specjalistyczny im sw. Jana Paw?a II, Krakow
  - Warminsko-Mazurskie Centrum Chorób P?uc w Olsztynie, Olsztyn
  - Wielkopolskie Centrum Pulmonologii i Torakochirurgii w Poznaniu, Poznan
- Romania (2):
  - Prof Dr I Chiricuta Institute of Oncology, Cluj-Napoca
  - Oncomed SRL, Timișoara
- Russia (7):
  - Moscow City Oncology Hospital #62, Moscovskaya Oblast, Moscow Oblast
  - FSBI Russian Oncology Research Center n.a. Blokhin of MOH RF, Moscow, Moscow Oblast
  - P.A. Gertsen Cancer Research Inst., Moscow, Moscow Oblast
  - Pavlov First Saint Petersburg State Medical University, Saint Petersburg, Sankt-Peterburg
  - SPb City Clin Onc Dsp, Saint Petersburg, Sankt-Peterburg
  - Scientific Research Oncology Institute named after N.N. Petrov, Saint Petersburg, Sankt-Peterburg
  - GUZ Regional clinical hospital # 1, Krasnodar
- South Korea (8):
  - National Cancer Center, Gyeonggi-do
  - Seoul National University Bundang Hospital, Gyeonggi-do
  - Ajou University Medical Center, Gyeonggi-do
  - Gachon University Gil Medical Center, Incheon
  - Chonnam National University Hwasun Hospital, Jeollanam-do
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
  - Korea University Guro Hospital, Seoul
- Spain (6):
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital Universitari Germans Trias i Pujol, Barcelona
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario Virgen del Rocio, Seville
  - Hospital Clinico Universitario de Valencia, Valencia
- Taiwan (5):
  - Chang Gung Memorial Foundation - Kaohsiung, Kaohsiung City
  - China Medical University Hospital, Taichung
  - National Taiwan University Hospital, Taipei
  - Chang Gung Medical Foundation - Linkou, Taoyuan District
  - Taichung Veterans General Hospital, Xitun Dist.
- Thailand (2):
  - Ramathibodi Hospital, Bangkok
  - Siriraj Hospital, Bangkok
- Turkey (Türkiye) (8):
  - Baskent University Adana Dr. Turgut Noyan Practice and Research Hospital, Adana
  - Hacettepe Uni Medical Faculty Hospital, Ankara
  - Ankara Ataturk Chest Diseases Training and Research Hospital, Ankara
  - Istanbul Uni Cerrahpasa Medical Faculty Hospital, Istanbul
  - Ege Uni Medical Faculty Hospital, Izmir
  - Izmir Suat Seren Chest Diseases and Surgery Research Hospital, Izmir
  - Inonu University Medical Faculty Turgut Ozal Medical Center Medical Oncology Department, Malatya
  - Medikal Park Samsun, Samsun
- Ukraine (5):
  - Medical center of Yuriy Spizhenko LLC, Kapitanovka Village, KIEV Governorate
  - Chemotherapy SI Dnipropetrovsk MA of MOHU, Dnipropetrovsk
  - Kyiv City Clinical Oncological Center, Kyiv
  - RCI Sumy Regional Clinical Oncological Dispensary, Sumy
  - Vinnytsia Regional Clinical Oncology Dispensary, Vinnytsia
- United Kingdom (2):
  - Guys Hospital, London
  - Wythenshaw Hospital, Manchester

IPD SHARING:
Plan to Share IPD: Yes
For eligible studies, qualified researchers may request access to individual patient level clinical data. See Roche's commitment to transparency of clinical study information here: https://go.roche.com/data_sharing

REFERENCES:
- [Derived] Wu YL, Dziadziuszko R, Ahn JS, Barlesi F, Nishio M, Lee DH, Lee JS, Zhong W, Horinouchi H, Mao W, Hochmair M, de Marinis F, Migliorino MR, Bondarenko I, Lu S, Wang Q, Lohmann TO, Xu T, Cardona A, Hiles L, Noe J, Solomon BJ. Plain language summary of the ALINA study results: alectinib compared with chemotherapy after surgery in people with ALK-positive non-small cell lung cancer. Future Sci OA. 2025 Dec;11(1):2578145. doi: 10.1080/20565623.2025.2578145. Epub 2025 Nov 11. PMID 41217067
- [Derived] Wu YL, Dziadziuszko R, Ahn JS, Barlesi F, Nishio M, Lee DH, Lee JS, Zhong W, Horinouchi H, Mao W, Hochmair M, de Marinis F, Migliorino MR, Bondarenko I, Lu S, Wang Q, Ochi Lohmann T, Xu T, Cardona A, Ruf T, Noe J, Solomon BJ; ALINA Investigators. Alectinib in Resected ALK-Positive Non-Small-Cell Lung Cancer. N Engl J Med. 2024 Apr 11;390(14):1265-1276. doi: 10.1056/NEJMoa2310532. PMID 38598794

RESULTS

PARTICIPANT FLOW:
Groups:
- Alectinib: Participants received 600 mg oral alectinib twice daily (BID) for 2 years
- Platinum-Based Chemotherapy: Participants received platinum-based chemotherapy for 4 cycles (cycle length = 21 days).
Period: Overall Study
Arm/Group | Alectinib | Platinum-Based Chemotherapy
Started | 130 | 127
Completed | 0 | 0
Not Completed | 130 | 127
Not completed — Withdrawal by Subject | 5 | 9
Not completed — Protocol deviation | 0 | 1
Not completed — Lost to Follow-up | 0 | 1
Not completed — Death | 2 | 5
Not completed — Study ongoing | 123 | 111

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Alectinib | Platinum-Based Chemotherapy | Total
Number analyzed (Participants) | 130 | 127 | 257
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.4 (12.5) | 56.6 (11.3) | 54.9 (12.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 75 | 59 | 134
  Male | 55 | 68 | 123
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 127 | 122 | 249
  Unknown or Not Reported | 2 | 5 | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 72 | 71 | 143
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 55 | 52 | 107
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 4 | 6

OUTCOME MEASURES:

1. Primary Outcome: Disease-free Survival (DFS), as Assessed by the Investigator
Description: DFS, defined as the time from randomization to the first documented recurrence of disease or new primary NSCLC as determined by the investigator through use of an integrated assessment of radiographic data, biopsy sample results (if clinically feasible), and clinical status or death from any cause, whichever occurs first
Time Frame: Approximately 58 months
Population: The ITT population consisted of all randomized participants, whether or not the participant received the assigned treatment.
  The Stage II-IIIa population consisted of all participants in the ITT population with Stage II-IIIa NSCLC.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Alectinib | Platinum-Based Chemotherapy
Number analyzed (Participants) | 15 | 50
months
  Stage II-IIIA population: number analyzed (Participants) | 14 | 45
  Stage II-IIIA population | NA [NA to NA] — The number of events is too low to estimate this parameter. | 44.4 [27.8 to NA] — There was insufficient follow-up time to estimate the upper limit.
  ITT population | NA [NA to NA] — The number of events is too low to estimate this parameter. | 41.3 [28.5 to NA] — There was insufficient follow-up time to estimate the upper limit.
Statistical Analysis 1: Comparison: Alectinib vs Platinum-Based Chemotherapy; Test type: Superiority; p = .0001, Log Rank; Hazard Ratio (HR) = 0.24, 95% CI 2-sided [0.13 to 0.45]
Statistical Analysis 2: Comparison: Alectinib vs Platinum-Based Chemotherapy; Test type: Superiority; p = .0001, Log Rank; Hazard Ratio (HR) = 0.24, 95% CI 2-sided [0.13 to 0.43]

2. Secondary Outcome: Overall Survival (OS)
Description: Primary OS analysis at approximately 5 years after FPI and final OS analysis at approximately 8 years after FPI.
  OS, defined as the time from randomization to death from any cause.
Time Frame: From the date of randomization until death due to any cause up to approximately 8 years
Reporting Status: Not Posted, anticipated posting 2026-11

3. Secondary Outcome: Percentage of Participants With Adverse Events (AEs)
Description: An adverse event is any untoward medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with the treatment. An adverse event can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a pharmaceutical product, whether or not considered related to the pharmaceutical product. Pre-existing conditions which worsen during a study are also considered as adverse events.
Time Frame: Until 28 days after the last dose of alectinib (up to 2 years) or 28 days after end of last cycle of chemotherapy (up to 4 cycles)
Population: The safety-evaluable population consisted of all participants who received at least one dose of study treatment, with participants assigned to treatment groups according to the treatment received. All participants who received any dose of alectinib are included in the alectinib treatment arm.
Measure: Number; unit: Percentage of participants
Arm/Group | Alectinib | Platinum-Based Chemotherapy
Number analyzed (Participants) | 128 | 120
Percentage of participants
  At least one AE | 98.4 | 93.3
  AE with fatal outcome | 0 | 0
  Grade 3-5 AE | 29.7 | 30.8
  Serious AE (SAE) | 13.3 | 8.3
  SAE leading to treatment withdrawal | 0.8 | 3.3
  SAE leading to dose modification/interruption | 5.5 | 3.3
  Related SAE | 1.6 | 6.7
  AE leading to treatment withdrawal | 5.5 | 12.5
  AE leading to dose modification/interruption | 43.0 | 22.5
  Related AE | 93.8 | 89.2
  Related AE leading to treatment withdrawal | 5.5 | 11.7
  Related AE leading to dose mod./interruption | 38.3 | 21.7

4. Secondary Outcome: AEs Grade 3-5 With a Difference in Incidence Rate of at Least 2% Between Treatment Arms
Description: as for outcome 3
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Number; unit: Percentage of participants
Arm/Group | Alectinib | Platinum-Based Chemotherapy
Number analyzed (Participants) | 128 | 120
Percentage of participants
  Neutrophil count decreased | 0 | 10.0
  Blood creatinine phosphokinase increased | 6.3 | 0.8
  White blood cell count decreased | 0 | 3.3
  Nausea | 0 | 4.2
  Appendicitis | 3.1 | 0
  Neutropenia | 0 | 8.3
  Asthenia | 0 | 2.5

5. Secondary Outcome: Plasma Concentration of Alectinib
Time Frame: Predose (2 hours) Week 3 - Week 96
Population: The PK-evaluable population consisted of all participants who received at least one dose of alectinib and who had at least one post-baseline PK sample available. This population did not include participants from the platinum-based chemotherapy arm, who did not receive alectinib.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Alectinib
Number analyzed (Participants) | 124
ng/mL
  Week 3: number analyzed (Participants) | 118
  Week 3 | 382 (276.2)
  Week 6: number analyzed (Participants) | 116
  Week 6 | 611 (70.6)
  Week 9: number analyzed (Participants) | 114
  Week 9 | 593 (91.4)
  Week 12: number analyzed (Participants) | 113
  Week 12 | 581 (94.9)
  Week 24: number analyzed (Participants) | 111
  Week 24 | 619 (93.2)
  Week 36: number analyzed (Participants) | 107
  Week 36 | 639 (54.1)
  Week 48: number analyzed (Participants) | 103
  Week 48 | 551 (90.1)
  Week 60: number analyzed (Participants) | 102
  Week 60 | 588 (58.9)
  Week 72: number analyzed (Participants) | 97
  Week 72 | 527 (96.5)
  Week 84: number analyzed (Participants) | 81
  Week 84 | 515 (91.1)
  Week 96: number analyzed (Participants) | 68
  Week 96 | 478 (106.4)

6. Secondary Outcome: Plasma Concentration of Alectinib Metabolite M4
Time Frame: Predose (2 hours) Week 3 - Week 96
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Alectinib
Number analyzed (Participants) | 124
ng/mL
  Week 3: number analyzed (Participants) | 119
  Week 3 | 178 (111.7)
  Week 6: number analyzed (Participants) | 119
  Week 6 | 214 (86.3)
  Week 9: number analyzed (Participants) | 116
  Week 9 | 213 (78.9)
  Week 12: number analyzed (Participants) | 115
  Week 12 | 205 (94.7)
  Week 24: number analyzed (Participants) | 111
  Week 24 | 237 (73.2)
  Week 36: number analyzed (Participants) | 107
  Week 36 | 238 (50.7)
  Week 48: number analyzed (Participants) | 102
  Week 48 | 209 (51.7)
  Week 60: number analyzed (Participants) | 102
  Week 60 | 217 (49.7)
  Week 72: number analyzed (Participants) | 97
  Week 72 | 213 (62.6)
  Week 84: number analyzed (Participants) | 81
  Week 84 | 198 (65.4)
  Week 96: number analyzed (Participants) | 68
  Week 96 | 191 (76.8)

ADVERSE EVENTS:
Time Frame: Until 28 days after the last dose of alectinib (up to 2 years) or 28 days after end of last cycle of chemotherapy (up to 4 cycles)
Description: All-cause mortality is reported for all participants.
  SAEs and Other AEs are reported for the safety-evaluable population, which consisted of all randomized participants who were enrolled during the global enrollment phase and received any amount of study drug, with participants grouped according to treatment received.
Arm/Group | Alectinib | Platinum-Based Chemotherapy
All-Cause Mortality (participants affected / at risk) | 2/130 | 5/127
Serious Adverse Events (participants affected / at risk) | 17/128 | 10/120
Other Adverse Events (participants affected / at risk) | 124/128 | 110/120
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Alectinib (N=128) | Platinum-Based Chemotherapy (N=120)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 2 (2) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Epigastric discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastritis erosive (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ileus paralytic (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 2 (2)
Pancreatitis acute (Gastrointestinal disorders) | 0 (0) | 1 (1)
Regurgitation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 0 (0) | 1 (1)
Appendicitis (Infections and infestations) | 4 (4) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 3 (3) | 1 (1)
Pneumonia viral (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Urosepsis (Infections and infestations) | 1 (1) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 2 (2)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Uterine prolapse (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Embolism (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Alectinib (N=128) | Platinum-Based Chemotherapy (N=120)
Anaemia (Blood and lymphatic system disorders) | 30 (45) | 31 (45)
Leukopenia (Blood and lymphatic system disorders) | 1 (1) | 9 (14)
Neutropenia (Blood and lymphatic system disorders) | 2 (2) | 19 (34)
Bradycardia (Cardiac disorders) | 10 (12) | 0 (0)
Constipation (Gastrointestinal disorders) | 54 (62) | 30 (34)
Diarrhoea (Gastrointestinal disorders) | 16 (17) | 10 (14)
Nausea (Gastrointestinal disorders) | 10 (12) | 87 (174)
Vomiting (Gastrointestinal disorders) | 9 (12) | 30 (62)
Asthenia (General disorders) | 14 (17) | 19 (29)
Fatigue (General disorders) | 18 (18) | 15 (21)
Malaise (General disorders) | 6 (6) | 16 (24)
Oedema peripheral (General disorders) | 13 (17) | 1 (1)
Pyrexia (General disorders) | 7 (9) | 4 (4)
COVID-19 (Infections and infestations) | 37 (38) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 9 (17) | 1 (1)
Urinary tract infection (Infections and infestations) | 11 (18) | 1 (2)
Alanine aminotransferase increased (Investigations) | 43 (60) | 11 (13)
Aspartate aminotransferase increased (Investigations) | 53 (77) | 6 (8)
Bilirubin conjugated increased (Investigations) | 11 (21) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 32 (48) | 4 (6)
Blood bilirubin increased (Investigations) | 43 (73) | 1 (1)
Blood creatine phosphokinase increased (Investigations) | 55 (74) | 1 (1)
Blood creatinine increased (Investigations) | 19 (26) | 6 (7)
Blood lactate dehydrogenase increased (Investigations) | 9 (13) | 6 (10)
Gamma-glutamyltransferase increased (Investigations) | 4 (4) | 7 (7)
Neutrophil count decreased (Investigations) | 3 (7) | 20 (48)
Platelet count decreased (Investigations) | 3 (4) | 6 (12)
Weight increased (Investigations) | 17 (25) | 1 (1)
White blood cell count decreased (Investigations) | 2 (4) | 23 (44)
Decreased appetite (Metabolism and nutrition disorders) | 7 (7) | 35 (53)
Hyperuricaemia (Metabolism and nutrition disorders) | 12 (21) | 2 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 10 (10) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 7 (7) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 36 (44) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 7 (7) | 2 (2)
Dizziness (Nervous system disorders) | 9 (10) | 11 (15)
Dysgeusia (Nervous system disorders) | 13 (18) | 3 (4)
Headache (Nervous system disorders) | 14 (15) | 8 (9)
Cough (Respiratory, thoracic and mediastinal disorders) | 19 (20) | 4 (4)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 13 (14) | 3 (3)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 9 (13)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 3 (3) | 7 (7)
Pruritus (Skin and subcutaneous tissue disorders) | 8 (8) | 3 (3)
Rash (Skin and subcutaneous tissue disorders) | 18 (21) | 7 (9)
Hypertension (Vascular disorders) | 4 (7) | 6 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2021-12-16): https://cdn.clinicaltrials.gov/large-docs/76/NCT03456076/Prot_000.pdf
  • Statistical Analysis Plan (2022-11-24): https://cdn.clinicaltrials.gov/large-docs/76/NCT03456076/SAP_001.pdf